CLINICAL TRIAL: NCT02712229
Title: A Cluster Randomized Trial of a Primary Palliative Care Intervention (CONNECT) for Patients With Advanced Cancer
Brief Title: A Primary Palliative Care Intervention for Patients With Advanced Cancer
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yael Schenker, MD, MAS, MD, MAS, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO15120154; 5R01CA197103-02 (NIH)
Record Dates: First submitted 2016-03-07; First posted 2016-03-18 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONNECT Intervention (Experimental): At clinics randomized to the CONNECT intervention, oncology nurses will be selected by a nurse advisory panel to receive standardized primary palliative care training. A multi-step deployment strategy will be employed to orient oncologists and implement CONNECT processes. CONNECT nurses will administer CONNECT to enrolled patients and caregivers. An intervention fidelity monitoring and maintenance plan will be implemented to ensure high quality and consistent delivery of the intervention.
  Interventions: Behavioral: CONNECT
- Usual Care Control (No Intervention): At clinics randomized to Usual Care, enrolled patients and caregivers will continue to receive supportive oncology care according to usual practice.

INTERVENTIONS:
Behavioral: CONNECT — Primary palliative care, care management intervention led by existing oncology nurses. Deployed through a series of nurse-led encounters before or after regularly scheduled oncology visits. Based on best practices in palliative oncology care, the first visit focuses on establishing rapport, addressing symptom needs and choosing a surrogate decision maker. Subsequent visits include additional focus on treatment preferences and future goals.
  Visits are guided by patient-reported outcomes. During all encounters, the nurse works with patients/caregivers to complete/update individualized Shared Care Plans. After all visits, the nurse discusses patients' symptoms, preferences and goals with their oncologists via a mandatory check-in session and a follow-up call with the patient and/or caregiver.
  Arms: CONNECT Intervention

SUMMARY:
The overall goal of this study is to test whether a nurse-led intervention to improve provision of primary palliative care within oncology practices (CONNECT) can decrease morbidity for patients with advanced cancer and their caregivers.

The specific aims are to:

Aim 1. Assess the effects of CONNECT on patient quality of life (primary outcome), symptom burden, and mood at 3-month follow-up.

Aim 2. Assess the effects of CONNECT on caregiver burden and mood at 3-month follow-up.

Aim 3. Assess the effects of CONNECT on healthcare resource use over 1 year of follow-up.

DETAILED DESCRIPTION:
Study investigators will conduct a cluster randomized controlled trial comparing the CONNECT intervention to usual care in 16 oncology clinics. CONNECT (Care Management by Oncology Nurses to address supportive care needs) is a care management intervention using existing oncology nurses to improve provision of primary palliative care within outpatient oncology practices.

The study will enroll 672 patients with advanced cancer and their caregivers. The study will assess the intervention's impact on patient and caregiver quality-of-life and psychological outcomes at three months and on healthcare utilization through one year of follow up. Investigators will follow a rigorous plan to establish and maintain intervention fidelity. Detailed process information will be collected at all sites and the study will evaluate how CONNECT impacts mortality and costs.

Following best practices for complex system-level interventions, the study will use a cluster randomized trial design. The unit of randomization is the oncology practice, defined as a unique location and provider group for outpatient oncology care. The unit of analysis is the individual patient and caregiver.

Designated staff at each clinic will review oncologists' schedules on a weekly basis to identify and track potentially eligible patients with an upcoming appointment. Research staff will review tracking systems weekly to maintain recruitment fidelity. Identified patients will receive a 1-page study information sheet at their next clinic visit, followed by a detailed in-person explanation of the study from a trained staff member. This staff member will obtain informed consent from all participants. To minimize potential selection bias, participants will be told in advance of both groups and not randomized if they decline to be exposed to one of them.

To enhance retention, blinded research assistants will conduct monthly follow-up calls to assess healthcare utilization for participants in both groups. The data collection strategy is designed to minimize participant burden by using parsimonious measures previously pilot-tested with this population.

ELIGIBILITY:
Participants will be (1) patients with advanced cancer receiving care at a participating clinic; (2) their caregivers; (3) their oncology staff nurses, oncologists, and practice managers.

Patient eligibility criteria. Inclusion criteria: (1) adults (≥ 21 years old); (2) the oncologist "would not be surprised if the patient died in the next year"; (3) Eastern Cooperative Oncology Group performance status (ECOG PS) of ≤ 2; (4) planning to receive ongoing care from a participating oncologist and willing to be seen at least monthly.

Exclusion criteria: (1) Unable to read and respond to questions in English; (2) cognitive impairment or inability to consent to treatment, as determined by the patient's oncologist; (3) unable to complete baseline interview; (4) ECOG PS of 3 (capable of limited self-care; confined to bed or chair > 50% of waking hours) or 4 (cannot carry on any self-care; totally confined to bed or chair); (5) hematologic malignancy.

Caregiver eligibility criteria. Inclusion criteria: (1) adults (≥ 21 years old); (2) family member or friend of an eligible patient. Exclusion criteria: (1) unable to read and respond to questions in English; (2) unable to complete the baseline interview. Patients will be asked to select as caregiver the person who is most likely to accompany them to visits or help with their care should they need it.

Clinician eligibility criteria. Oncology staff nurses who undergo training to deploy CONNECT, oncologists, and practice managers at participating sites will be eligible to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1290 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Quality of Life - patient | Change from baseline to 3 months
  The investigators will compare change in the 3-month FACIT-Pal scores between enrolled patients at intervention clinics and enrolled patients at usual care clinics.

SECONDARY OUTCOMES:
Symptom burden - patient | Change from baseline to 3 months
  The investigators will compare change in the 3-month Edmonton Symptom Assessment Scale (ESAS) scores between enrolled patients at intervention clinics and enrolled patients at usual care clinics.
Depression and anxiety symptoms - patient | Change from baseline to 3 months
  The investigators will compare change in the 3-month Hospital Anxiety and Depression Scale (HADS) scores between enrolled patients at intervention clinics and enrolled patients at usual care clinics.
Depression and anxiety symptoms - caregiver | Change from baseline to 3 months
  The investigators will compare change in the 3-month Hospital Anxiety and Depression Scale (HADS) scores between enrolled caregivers at intervention clinics and enrolled caregivers at usual care clinics.
Caregiver burden - caregiver | Change from baseline to 3 months
  The investigators will compare change in the 3-month Zarit Burden Interview-Short scores between enrolled caregivers at intervention clinics and enrolled caregivers at usual care clinics.
Healthcare Utilization | 1 year
  To inform future dissemination efforts and aid in understanding optimal financing models, the investigators will calculate implementation costs of the intervention and determine the effects of CONNECT on healthcare utilization, including hospitalizations, chemotherapy use, and hospice use.
Survival - patients | 1 year
  The investigators will calculate survival time from date of enrollment using the Kaplan-Meier method. We will use frailty models to assess for any effect of CONNECT on survival, controlling for the effects of clustering.

OTHER OUTCOMES:
Patient-Oncologist Therapeutic Relationship | Change from baseline to 3 months
  The investigators will compare change in the 3-month Human Connection Scale scores between enrolled patients at intervention clinics and enrolled patients at usual care clinics.
Hope - patients and caregivers | Change from baseline to 3 months
  The investigators will compare change in the 3-month Herth Hope Index scores between enrolled patients and caregivers at intervention clinics and enrolled patients and caregivers at usual care clinics.
Self-efficacy - patients and caregivers | 3 months
  The investigators will compare 3-month scores on the Cancer Behavior Inventory-Brief (patients) and the Caregiver Inventory (caregivers) between enrolled patients and caregivers at intervention clinics and enrolled patients and caregivers at usual care clinics.
Satisfaction - caregivers | Change from baseline to 3 months
  The investigators will compare change in the 3-month FAMCARE-2 scores between enrolled caregivers at intervention clinics and enrolled caregivers at usual care clinics.
Distress - patients | Change from baseline to 3 months
  The investigators will compare change in the 3 months scores on the Distress Thermometer between enrolled patients at intervention clinics and enrolled patients at usual care clinics.
Illness understanding, care preferences, advance care planning - patients | Change from baseline to 3 months
  The investigators will compare change in patient illness understanding, care preferences, and advance care planning between enrolled patients at intervention clinics and enrolled patients at usual care clinics.
Burnout - clinicians | Baseline and annually up to 60 months
  The investigators will compare burnout (maslach burnout inventory) between clinicians at intervention clinics and usual care clinics.
Satisfaction with CONNECT and recommendations for improvement | Annually up to 60 months
  The investigators will assess satisfaction with CONNECT and recommendations for improvement among clinicians at intervention clinics annually.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Schenker, MD, MAS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schenker Y, White D, Rosenzweig M, Chu E, Moore C, Ellis P, Nikolajski P, Ford C, Tiver G, McCarthy L, Arnold R. Care management by oncology nurses to address palliative care needs: a pilot trial to assess feasibility, acceptability, and perceived effectiveness of the CONNECT intervention. J Palliat Med. 2015 Mar;18(3):232-40. doi: 10.1089/jpm.2014.0325. Epub 2014 Dec 17. PMID 25517219
- [Background] Downey L, Engelberg RA. Quality-of-life trajectories at the end of life: assessments over time by patients with and without cancer. J Am Geriatr Soc. 2010 Mar;58(3):472-9. doi: 10.1111/j.1532-5415.2010.02734.x. PMID 20398115
- [Background] Giesinger JM, Wintner LM, Oberguggenberger AS, Gamper EM, Fiegl M, Denz H, Kemmler G, Zabernigg A, Holzner B. Quality of life trajectory in patients with advanced cancer during the last year of life. J Palliat Med. 2011 Aug;14(8):904-12. doi: 10.1089/jpm.2011.0086. Epub 2011 Jun 28. PMID 21711125
- [Background] Zhang B, Wright AA, Huskamp HA, Nilsson ME, Maciejewski ML, Earle CC, Block SD, Maciejewski PK, Prigerson HG. Health care costs in the last week of life: associations with end-of-life conversations. Arch Intern Med. 2009 Mar 9;169(5):480-8. doi: 10.1001/archinternmed.2008.587. PMID 19273778
- [Background] Wright AA, Zhang B, Ray A, Mack JW, Trice E, Balboni T, Mitchell SL, Jackson VA, Block SD, Maciejewski PK, Prigerson HG. Associations between end-of-life discussions, patient mental health, medical care near death, and caregiver bereavement adjustment. JAMA. 2008 Oct 8;300(14):1665-73. doi: 10.1001/jama.300.14.1665. PMID 18840840
- [Background] Barnato AE, Herndon MB, Anthony DL, Gallagher PM, Skinner JS, Bynum JP, Fisher ES. Are regional variations in end-of-life care intensity explained by patient preferences?: A Study of the US Medicare Population. Med Care. 2007 May;45(5):386-93. doi: 10.1097/01.mlr.0000255248.79308.41. PMID 17446824
- [Background] Northouse LL, Katapodi MC, Schafenacker AM, Weiss D. The impact of caregiving on the psychological well-being of family caregivers and cancer patients. Semin Oncol Nurs. 2012 Nov;28(4):236-45. doi: 10.1016/j.soncn.2012.09.006. PMID 23107181
- [Background] Detmar SB, Aaronson NK, Wever LD, Muller M, Schornagel JH. How are you feeling? Who wants to know? Patients' and oncologists' preferences for discussing health-related quality-of-life issues. J Clin Oncol. 2000 Sep 15;18(18):3295-301. doi: 10.1200/JCO.2000.18.18.3295. PMID 10986063
- [Background] Detmar SB, Muller MJ, Wever LD, Schornagel JH, Aaronson NK. The patient-physician relationship. Patient-physician communication during outpatient palliative treatment visits: an observational study. JAMA. 2001 Mar 14;285(10):1351-7. doi: 10.1001/jama.285.10.1351. PMID 11255393
- [Background] Pollak KI, Arnold RM, Jeffreys AS, Alexander SC, Olsen MK, Abernethy AP, Sugg Skinner C, Rodriguez KL, Tulsky JA. Oncologist communication about emotion during visits with patients with advanced cancer. J Clin Oncol. 2007 Dec 20;25(36):5748-52. doi: 10.1200/JCO.2007.12.4180. PMID 18089870
- [Background] Temel JS, Greer JA, Admane S, Solis J, Cashavelly BJ, Doherty S, Heist R, Pirl WF. Code status documentation in the outpatient electronic medical records of patients with metastatic cancer. J Gen Intern Med. 2010 Feb;25(2):150-3. doi: 10.1007/s11606-009-1161-z. Epub 2009 Nov 6. PMID 19894078
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Bakitas M, Lyons KD, Hegel MT, Balan S, Brokaw FC, Seville J, Hull JG, Li Z, Tosteson TD, Byock IR, Ahles TA. Effects of a palliative care intervention on clinical outcomes in patients with advanced cancer: the Project ENABLE II randomized controlled trial. JAMA. 2009 Aug 19;302(7):741-9. doi: 10.1001/jama.2009.1198. PMID 19690306
- [Background] Zimmermann C, Swami N, Krzyzanowska M, Hannon B, Leighl N, Oza A, Moore M, Rydall A, Rodin G, Tannock I, Donner A, Lo C. Early palliative care for patients with advanced cancer: a cluster-randomised controlled trial. Lancet. 2014 May 17;383(9930):1721-30. doi: 10.1016/S0140-6736(13)62416-2. Epub 2014 Feb 19. PMID 24559581
- [Background] Hui D, Elsayem A, De la Cruz M, Berger A, Zhukovsky DS, Palla S, Evans A, Fadul N, Palmer JL, Bruera E. Availability and integration of palliative care at US cancer centers. JAMA. 2010 Mar 17;303(11):1054-61. doi: 10.1001/jama.2010.258. PMID 20233823
- [Background] Maciasz RM, Arnold RM, Chu E, Park SY, White DB, Vater LB, Schenker Y. Does it matter what you call it? A randomized trial of language used to describe palliative care services. Support Care Cancer. 2013 Dec;21(12):3411-9. doi: 10.1007/s00520-013-1919-z. Epub 2013 Aug 14. PMID 23942596
- [Background] Schenker Y, Park SY, Maciasz R, Arnold RM. Do patients with advanced cancer and unmet palliative care needs have an interest in receiving palliative care services? J Palliat Med. 2014 Jun;17(6):667-72. doi: 10.1089/jpm.2013.0537. Epub 2014 Mar 27. PMID 24673544
- [Background] Schenker Y, Crowley-Matoka M, Dohan D, Rabow MW, Smith CB, White DB, Chu E, Tiver GA, Einhorn S, Arnold RM. Oncologist factors that influence referrals to subspecialty palliative care clinics. J Oncol Pract. 2014 Mar;10(2):e37-44. doi: 10.1200/JOP.2013.001130. Epub 2013 Dec 3. PMID 24301842
- [Derived] Booth G, Rahman M, Rosenzweig M, Thomas TH, Schenker Y. What's on your mind? A qualitative analysis of concerns and self-management strategies among older adults with advanced cancer. J Geriatr Oncol. 2025 Sep;16(7):102328. doi: 10.1016/j.jgo.2025.102328. Epub 2025 Aug 8. PMID 40782786
- [Derived] Bell SG, Althouse AD, Belin SC, Arnold RM, Smith KJ, White DB, Chu E, Schenker Y, Thomas TH. Associations of Health Care Utilization and Therapeutic Alliance in Patients with Advanced Cancer. J Palliat Med. 2024 Apr;27(4):515-520. doi: 10.1089/jpm.2023.0559. PMID 38574330
- [Derived] Mitchell CJ, Althouse A, Feldman R, Arnold RM, Rosenzweig M, Smith K, Chu E, White D, Smith T, Schenker Y. Symptom Burden and Shared Care Planning in an Oncology Nurse-Led Primary Palliative Care Intervention (CONNECT) for Patients with Advanced Cancer. J Palliat Med. 2023 May;26(5):667-673. doi: 10.1089/jpm.2022.0277. Epub 2022 Dec 5. PMID 36472545
- [Derived] Sigler LE, Althouse AD, Thomas TH, Arnold RM, White D, Smith TJ, Chu E, Rosenzweig M, Smith KJ, Schenker Y. Effects of an Oncology Nurse-Led, Primary Palliative Care Intervention (CONNECT) on Illness Expectations Among Patients With Advanced Cancer. JCO Oncol Pract. 2022 Apr;18(4):e504-e515. doi: 10.1200/OP.21.00573. Epub 2021 Nov 12. PMID 34767474
- [Derived] Schenker Y, Althouse AD, Rosenzweig M, White DB, Chu E, Smith KJ, Resick JM, Belin S, Park SY, Smith TJ, Bakitas MA, Arnold RM. Effect of an Oncology Nurse-Led Primary Palliative Care Intervention on Patients With Advanced Cancer: The CONNECT Cluster Randomized Clinical Trial. JAMA Intern Med. 2021 Nov 1;181(11):1451-1460. doi: 10.1001/jamainternmed.2021.5185. PMID 34515737
- [Derived] Thomas T, Althouse A, Sigler L, Arnold R, Chu E, White DB, Rosenzweig M, Smith K, Smith TJ, Schenker Y. Stronger therapeutic alliance is associated with better quality of life among patients with advanced cancer. Psychooncology. 2021 Jul;30(7):1086-1094. doi: 10.1002/pon.5648. Epub 2021 Mar 8. PMID 33547717

DOCUMENTS (1):
  • Informed Consent Form (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT02712229/ICF_000.pdf